CLINICAL TRIAL: NCT02541084
Title: Caregiver Burden of Wet Age-related Macular Degeneration (wAMD) Treatment in Real-life Japanese Settings.
Brief Title: Caregiver Burden of Wet Age-related Macular Degeneration (wAMD) in Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 17945
Record Dates: First submitted 2015-08-05; First posted 2015-09-04 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Wet Macular Degeneration
Keywords: Age-related macular degeneration; Caregiver burden; Anti-vascular endothelial growth factor (VEGF) therapy
MeSH Terms: conditions — Wet Macular Degeneration; Macular Degeneration; Caregiver Burden | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PRN group: wAMD-patients treated with anti-VEGF therapy ´pro re nata´ (PRN)
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- TAE group: wAMD-patients treated with anti-VEGF therapy ´treat-and-extend´ (TAE)
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)
- PRN-to-TAE switcher group: wAMD patients treated with anti-VEGF therapy and switching from PRN to TAE regimens
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Anti-VEGF therapy following the Summary of Product Characteristics

SUMMARY:
This study aims at investigation of the caregiver burden of Wet Age-related Macular Degeneration (wAMD) patients and at the assessment of how much of caregiver burden could be reduced in transitioning from Pro Re Nata to proactive therapy especially in real-life rural settings where public transportations are not readily available.

ELIGIBILITY:
Inclusion Criteria:

* [Patients]

  * Female and male out-patients diagnosed with wAMD.
  * Patients who are accompanied by his/her caregiver(s).
  * Patients who have been receiving anti-VEGF therapy with proactive regimen for 12 months or more at the participating site.
  * Providing informed consent for the participation in this study.
* [Caregivers]

  * Providing informed consent for the participation in this study.
  * Capable of understanding and completing the questionnaires without any help from others

Exclusion Criteria:

* [Patients]

  * Presence of a disease or a condition more disabling than wAMD in term of caregiving.
  * Presence of intractable neurologic disease, physical handicap, mental handicap, or any condition that rendered them unable to walk independently.
  * Intraocular surgery for other eye diseases after the start of wAMD therapy.
* [Caregivers]

  * Professional carers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Information on patients will be collected from all female and male out-patients with a diagnosis of wAMD who currently receive anti-VEGF therapy with proactive regimen at Kozawa Eye Hospital (Mito-city, Japan). Of these, patients who are accompanied by his/her caregiver and the caregiver (a pair of patient-caregiver) who satisfy eligibility listed below will be recruited for the assessment of primary and secondary objectives.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-08-18 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Degree of caregiving burden on caregivers (BIC-11) | At enrollment
  Burden Index of Caregivers (BIC), a multidimensional short care burden scale from Japan.The score range is from 0-40, with high scores indicating greater care giver burden.
Relationship between BIC-11 and the number of hospital visits for wAMD treatments | Up to 1 year
Frequency of hospital visits | Up to 1 year
Time spent by accompanying caregivers for a clinic visit for wAMD management (minutes) | Up to 1 year
Estimated costs spent by accompanying caregivers on hospital visits for wAMD management | Up to 1 year

SECONDARY OUTCOMES:
Level of depression among caregivers (CES-D) | At Enrollment
  CES-D will be applied to determine depression.The score range is from 0 to 60, with high score indicating greater depressive symptoms. Cut off score is 16 or greater in Japan to assess whether individuals experience depression.
Types of treatments for wAMD | At Baseline
  Anti-VEGF(anti vascular endothelial growth factor)drugs, laser therapy, Photodynamic Therapy,etc.
Frequency of treatments | At baseline
  Number of a therapeutic agent given to patients
Length of treatment | At baseline
  Duration of a therapeutic agent received
Dosing schedule | At baseline
  The schedule of doses of a therapeutic agent per unit of time
Percentage of patients accompanied by primary caregivers | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan